CLINICAL TRIAL: NCT04994795
Title: Deep Learning-Enabled Exploration of Predictive Signatures in a Multicenter Retrospective and Prospective Observational Study Allowing the Analysis of the Aggregation of Multimodal Clinical, Biological, Genomic and Radiomics Data Associated With the Response to Treatment and Prognosis of Patients With Stage IV Non-small Cell Lung Cancer
Brief Title: Predictive Multimodal Signatures Associated With Response to Treatment and Prognosis of Patients With Stage IV Non-small Cell Lung Cancer
Acronym: DEEP-Lung-IV
Status: Active, not recruiting | Type: Observational
Sponsor: Sophia Genetics SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: SGDLIV
Record Dates: First submitted 2021-07-15; First posted 2021-08-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: NSCLC; Immunotherapy; Chemotherapy; Predictive models; Radiomics; Multimodal; Genomics; Machine learning
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pembrolizumab monotherapy
  Interventions: Other: Predictive models (data collection)
- Chemotherapy and pembrolizumab combination therapy
  Interventions: Other: Predictive models (data collection)
- Chemotherapy doublet
  Interventions: Other: Predictive models (data collection)

INTERVENTIONS:
Other: Predictive models (data collection) — Machine learning predictive models

SUMMARY:
Predicting response to therapy and disease progression in stage IV NSCLC patients treated with pembrolizumab monotherapy, chemotherapy-pembrolizumab combination therapy or chemotherapy alone in the first-line setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years old
* Patient diagnosed with Stage IV NSCLC (de novo or earlier stage progression to stage IV)
* Absence of oncogene activating mutations eligible patients to targeted therapy (EGFR, ALK)
* Cohort A: Received first line treatment with pembrolizumab monotherapy
* Cohort B: Received first line treatment with chemotherapy and pembrolizumab combination therapy
* Cohort C: Received first line treatment with chemotherapy doublet

Exclusion Criteria:

* Prior anti-cancer therapy for actual stage IV NSCLC
* Critical data missing (e.g., PD-L1 status, baseline millimetric imaging, first evaluation millimetric imaging)
* Patients participating in other clinical trials that modify the standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with stage IV NSCLC (de novo or earlier stage progression to stage IV), without oncogene-activating mutations eligible for targeted therapy, that are treated in the first-line setting with either pembrolizumab monotherapy, chemotherapy and pembrolizumab combination therapy, or chemotherapy.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Treatment response at first evaluation | 6-12 weeks after treatment start
  Predict treatment response at first evaluation using baseline data

SECONDARY OUTCOMES:
Progression-Free Survival | Through study completion, expected 6-14 months contingent on cohort
  Predict Progression-Free Survival (PFS) using data at baseline and first evaluation
Overall Survival | Through study completion, expected 8-20 months contingent on cohort
  Predict Overall Survival (OS) using data at baseline and first evaluation
Duration of Response | Through study completion, expected 6-14 months contingent on cohort
  Predict Duration of Response (DoR) using data at baseline and first evaluation
Time-To-Progression | Through study completion, expected 6-14 months contingent on cohort
  Predict Time-To-Progression (TTP) using data at baseline and first evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Menu, MD-PhD, MBA, Study Director — SOPHiA GENETICS
Locations (30):
- United States (6):
  - Holden Comprehensive Cancer Center at University of Iowa Health Care, Iowa City, Iowa
  - UMASS Memorial Health, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Carbone Comprehensive Cancer Center at University of Wisconsin, Madison, Wisconsin
- Brazil (5):
  - DASA - Hospital Brasilia, Brasília
  - DASA - Hospital de Niteroi, Niterói
  - DASA - Hospital São Lucas, Rio de Janeiro
  - DASA - Hospital Nove De Julho, São Paulo
  - AC Camargo, São Paulo
- Sunnybrook Health Sciences Centre Toronto, Toronto, Canada
- France (9):
  - Avicenne Hospital, Bobigny
  - CHU Bordeaux, Bordeaux
  - Ambroise Paré Hospital, Boulogne-Billancourt
  - Hospices Civils de Lyon, Lyon
  - CHU de Nantes, Nantes
  - La Pitié Salpêtrière, Paris
  - Tenon Hospital, Paris
  - Foch Hospital, Suresnes
  - Centre Hospitalier de Toulon, Toulon
- University Hospital Leipzig, Leipzig, Germany
- Israel (2):
  - Shaare Zadek Medical Center, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (3):
  - University Hospital Of Parma, Parma
  - Policlinico Gemelli, Roma
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), Udine
- Spain (3):
  - Fundacion jimenez diaz, Madrid
  - Puerta De Hierro Hospital, Madrid
  - Instituto Valenciano De Oncologia, Valencia